CLINICAL TRIAL: NCT05676372
Title: The Role of the Peritoneal Microenvironment in the Pathogenesis of Colorectal Peritoneal Carcinomatosis: Single-cell Transcriptomics
Brief Title: Single-Cell Transcriptomics of the Peritoneal Microenvironment of Colorectal PC
Acronym: SingleCell
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Collaborators: Flemish institute of biotechnology (VIB) (Other)
Responsible Party: Sponsor
Other Study IDs: BC-6978
Record Dates: First submitted 2020-11-26; First posted 2023-01-09 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Peritoneal Metastases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peritoneal metastases (surgical waste material)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CRC+HIPEC — Sample prelevation of cytoreductive surgery

SUMMARY:
Single cell transcriptomics of CRC PC samples

DETAILED DESCRIPTION:
Research methodology

Before inclusion of patients, patients will be screened for the presence of hepatitis B, hepatitis C and HIV to ensure researcher safety. During cytoreductive surgery, a total of five samples of tumoral tissue will be acquired. Three of those samples will be utilized for ScRNASeq analysis, and two samples of a macrometastasis will be snap frozen and cryopreserved.

Single-cell RNA-Sequencing analysis We will comprehensively catalog the stromal cell types in the microenvironment of colorectal cancer peritoneal metastases utilizing single-cell RNA sequencing (scRNAseq) on three samples (one of which should preferably originate from the omentum majus, to encompass milky spots) acquired from surgical waste material of patients undergoing cytoreductive surgery. After sample prelevation, samples will be transported as soon as possible while cooled and submerged in 10% PBS to the VIB facilities, where single cell suspensions will be made according to standard protocols. After cell selection by FACS (CD45+ and live/dead stain, to ensure a 50/50 mix of immune and stromal cells) and library prep, ScRNASeq will be performed.

Single cell sequencing analysis will allow us to identify cell clusters that by usage of marker genes will be assigned to different known cell lineages. After annotation of data, a "landscape" of the composition of the tumor stroma will be acquired.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CRS+HIPEC for PC of colorectal origin

Exclusion Criteria:

* Previous HIPEC/PIPAC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing CRS+HIPEC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Single-cell transcriptomics | 24 months
  A transcriptional single-cell RNA seq atlas of gene expression data will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Wim Ceelen, MD, PhD, Principal Investigator — UZ Ghent
Locations (1):
- UZ Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No